CLINICAL TRIAL: NCT06326788
Title: Effects of Moderate Intensity Soleus Push-ups vs Sustained Soleus Push-ups on Lipid Profile Among Young Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3912 Mehnoor Butt
Record Dates: First submitted 2024-03-04; First posted 2024-03-22 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Health Behavior
Keywords: lipid profile; Young Population; Push-ups; Soleus; Sustained
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Duration Moderate Intensity Soleus Push-ups (Group A) (Experimental): Moderate physical activity involving weighted soleus push-ups performed till patient MHR is achieved.
  Interventions: Behavioral: Short Duration Moderate Intensity Soleus Push-ups
- Sustained Soleus Push-ups (Group B) (Experimental): sustained soleus push-ups will be performed for up to 270 min.
  Interventions: Behavioral: SUSTAINED SOLEUS PUSH-UPS

INTERVENTIONS:
Behavioral: Short Duration Moderate Intensity Soleus Push-ups — Participants will start soleus pushups in sitting positions. To do so, the participants will be in a seated position, the legs will be at 90 degrees to the floor, and the feet will be placed flat on the ground.
  Participants will then move their heels up and down continuously. Soleus push-ups will be performed with moderate intensity using weights which will be placed on their laps.
  Participants will perform this activity till 60-70% of their maximum heart rate is achieved and maintained.
  Other Names: Group A
  Arms: Short Duration Moderate Intensity Soleus Push-ups (Group A)
Behavioral: SUSTAINED SOLEUS PUSH-UPS — Participants will start soles push-ups in sitting. To do so, the participants will be in a seated position, the legs will be at 90 degrees to the floor, and the feet will be placed flat on the ground.
  Participants will then move their heels up and down continuously. Sustained soleus push-ups will be performed with light intensity for up to 270 mins.
  No external resistance will be added. Participants will be provided with a maximum 4-minute break time after every 90 mins intervention. In the meantime, their blood sample will be collected.
  Other Names: Group B
  Arms: Sustained Soleus Push-ups (Group B)

SUMMARY:
To determine the effects of Short duration moderate intensity soleus push- ups VS Sustained Soleus Push-ups on lipid profile among Young Population.

DETAILED DESCRIPTION:
The soleus muscle is a special type of muscle in our body that uses blood glucose for energy. It can work for a long time without getting tired. This muscle does not store energy like other muscles do. Instead, it directly uses the glucose in our blood.

Soleus push-ups are a type of exercise that targets this muscle. They could be really useful to stimulate our metabolism and keep blood lipids under control. Some studies suggest that doing soleus push-ups for a long time can positively affect our blood.

But we're not sure how different types of soleus pushups affect our blood fats. That's what this study wants to discover. We want to compare how doing sustained soleus curls for a long time compares to doing shorter, moderate intensity soleus curls. We want to see if the shorter ones can give us similar or even better results in improving our blood fats.

By conducting this study, we hope to learn more about how specific exercises can help us keep our hearts healthy and blood fats in balance. We will take a close look at the data we collect and use it to understand what type of exercise might be best for improving our blood fat levels.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age range: 18-26 )
* BMI: Healthy Young Adults.
* Equal number of gender
* Healthy young Adults.

Exclusion Criteria:

* History of metabolic diseases.
* History of recent fractures.
* Patient with any lower limb injuries.
* Knee injuries. The patient is already involved in regular physical exercise and a prescribed diet.
* Any deformity from childhood
* DVT and lower limb amputation.
* Known case of hyperlipidemia.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-07-28 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Lipid Profile | baseline to 6 hours
  The primary outcome measure will be the change in lipid profile parameters, including total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides, measured before and after the intervention period. This will provide insight into the direct impact of short duration moderate intensity Soleus push-ups vs sustained Soleus push-ups on lipid metabolism among young individuals.

OTHER OUTCOMES:
Adherence to Exercise Protocol | baseline to 6 hours
  Adherence to the prescribed exercise protocols, including the frequency, duration, and intensity of push-up sessions, will be monitored throughout the intervention period to assess compliance and determine if there are any differences in adherence between the two exercise groups.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Durstine JL, Grandjean PW, Cox CA, Thompson PD. Lipids, lipoproteins, and exercise. J Cardiopulm Rehabil. 2002 Nov-Dec;22(6):385-98. doi: 10.1097/00008483-200211000-00002. PMID 12464825
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Background] Holten MK, Zacho M, Gaster M, Juel C, Wojtaszewski JF, Dela F. Strength training increases insulin-mediated glucose uptake, GLUT4 content, and insulin signaling in skeletal muscle in patients with type 2 diabetes. Diabetes. 2004 Feb;53(2):294-305. doi: 10.2337/diabetes.53.2.294. PMID 14747278
- [Background] Swain DP, Franklin BA. Comparison of cardioprotective benefits of vigorous versus moderate intensity aerobic exercise. Am J Cardiol. 2006 Jan 1;97(1):141-7. doi: 10.1016/j.amjcard.2005.07.130. Epub 2005 Nov 16. PMID 16377300
- [Background] Taube W, Kullmann N, Leukel C, Kurz O, Amtage F, Gollhofer A. Differential reflex adaptations following sensorimotor and strength training in young elite athletes. Int J Sports Med. 2007 Dec;28(12):999-1005. doi: 10.1055/s-2007-964996. Epub 2007 May 11. PMID 17497570